CLINICAL TRIAL: NCT06823232
Title: A Study on the Substance Balance of [14C]XY0206 in Healthy Adult Chinese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: XY0206AML1006
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Metabolism of Radioactive Substances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C]XY0206 (Experimental): 37.5 mg/100 µCi [14C]XY0206
  Interventions: Drug: [14C]XY0206

INTERVENTIONS:
Drug: [14C]XY0206 — On the morning of the day of medication (D1), the subject took [14C] XY0206 suspension orally on an empty stomach (containing approximately 37.5 mg/100 µ Ci [14C] XY0206).

SUMMARY:
The main purpose of this clinical trial is to quantitatively analyse the total radioactivity in the excreta of subjects after oral administration of [14C]XY0206, and to obtain data on human radioactive excretion rate and main excretion routes and the radioactivity of human plasma, urine, and faeces after oral administration of [14C]XY0206 by subjects Metabolite profiling, identification of major metabolites, determination of metabolic pathways and elimination pathways; Subjects who met the criteria fasted for at least 10h before administration and took [14C]XY0206 suspension (containing about 37.5mg/100µCi[14C]XY0206) orally on an empty stomach in the morning of the first day of administration (DI).Subjects will also complete urine, stool and blood collection within a specified period of time。

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males;
2. Age: 18-45 years old (including boundary values);
3. Weight: The subject's weight is not less than 50 kg, and their body mass index (BMI) is between 19-26 kg/m2 (including boundary values);
4. Voluntary signing of informed consent form; The subjects are able to communicate well with the researchers and complete the experiment according to the protocol.

Exclusion Criteria:

* Supplementary Examination:

  1. Individuals who have undergone comprehensive physical examination, vital signs, routine laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, stool routine+occult blood), thyroid function, chest X-ray, abdominal ultrasound (liver, gallbladder, pancreas, spleen and kidney), and other examinations that are abnormal and clinically significant;
  2. Patients with clinically significant abnormal 12 lead electrocardiogram during the screening/baseline period, or those with QTc interval (QTcF) ≥ 450 ms corrected according to Fridericia's criteria;
  3. Individuals who are positive for any one of hepatitis B virus surface antigen, hepatitis B virus e antigen, hepatitis B virus core antibody, hepatitis C virus antibody, HIV antibody, and Treponema pallidum antibody.

     Medication history:
  4. Have used any drugs that inhibit or induce liver drug metabolizing enzymes within 28 days prior to administration (see Appendix 1 for details);
  5. Any medication that may cause QTc interval prolongation has been used within 28 days prior to administration (see Appendix 2 for details);
  6. Have used any prescription, over-the-counter, herbal or health supplements within 14 days prior to administration;
  7. Individuals who have participated in any clinical trials and received intervention with investigational drugs or medical devices within the last 3 months prior to the screening period;
  8. Screening individuals who have received the vaccine within the previous month or have a vaccination plan during the trial period;

History of illness and surgery:

9) Any clinical history of serious diseases or conditions that researchers believe may affect the test results, including but not limited to a history of motor system, nervous system, endocrine system, circulatory system, respiratory system, digestive system, urinary system, reproductive system diseases; 10) History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, twisted ventricular tachycardia, ventricular tachycardia, atrioventricular block, and any type of cardiovascular disease/disease/surgery that may increase QT interval prolongation, or a history of other risk factors leading to TdP (such as hypokalemia, hypomagnesemia, congenital long QT syndrome or family history of long QT syndrome or Brugada syndrome); 11) Having undergone major surgery or incomplete healing of surgical incision within the 6 months prior to the screening period; Major surgeries include but are not limited to any surgery involving significant bleeding risks, prolonged general anesthesia, or open biopsy or significant traumatic injuries; 12) Allergic constitution, such as those with a known history of allergies to two or more substances; Or those who may be allergic to the investigational drug or its excipients, as determined by researchers; 13) Clinically significant gastrointestinal abnormalities that may affect drug intake, transport, or absorption (such as inability to swallow, intestinal obstruction, digestive ulcers, etc.); Hemorrhoids or perianal diseases with regular/ongoing rectal bleeding, irritable bowel syndrome, inflammatory bowel disease; habits and customs: 15) Habitual constipation or diarrhea; 16) Excessive drinking or frequent alcohol consumption within the first 6 months of the screening period, i.e. drinking more than 14 units of alcohol per week (1 unit=360 mL of beer or 45 mL of 40% spirits or 150 mL of wine); 17) Individuals who smoke more than 5 cigarettes per day or habitually use nicotine containing products during the first 3 months of the screening period and are unable to quit during the trial period; 18) Individuals with a history of drug abuse or addiction in the past 5 years; 19) Habitual consumption of grapefruit juice or excessive amounts of tea, coffee, and/or caffeinated beverages, and inability to quit during the trial period; other: 20) Individuals with positive results in urine drug abuse screening and alcohol breath test during the baseline period; 21) Engage in work that requires long-term exposure to radioactive conditions; Or those who have had significant radiation exposure (≥ 2 chest/abdominal CT scans, or ≥ 3 other types of X-ray examinations) or have participated in radiopharmaceutical labeling trials within 1 year prior to the experiment; 22) Individuals with a history of needle or blood dizziness, difficulty in blood collection, or intolerance to venipuncture blood collection; 23) Those who have planned to give birth or donate sperm during the trial period and within 6 months after completion of the trial, or those who do not agree that the subjects and their spouses should take strict contraceptive measures during the trial period and within 6 months after completion of the trial; 24)Individuals who have experienced blood loss or donated up to 400 mL of blood within the past 3 months prior to the screening period, or who have received blood transfusions within the past 1 month; 25)Researchers believe that subjects with any factors that are not suitable for participation in this experiment

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
excrement | 22 days
  The total radioactivity of the collected biological samples (urine+feces) from each subject exceeds 90% of the administered dose, and the radioactivity collected for two consecutive days is less than 1% of the administered dose.
Radioactive blood sample | 22 days
  The total radioactive concentration of plasma samples is less than 3 times the background value

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Gaobo Hospital, Life Science Park Road, Changping District, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No